CLINICAL TRIAL: NCT03292042
Title: Impact of a Physical Health Promotion Program for People With Serious Mental Illness
Brief Title: Effectiveness of a Lifestyle Intervention, for People With SMI Who Meet Metabolic Syndrome Criteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 109-17
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2017-09

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; lifestyle intervention; health promotion; mental health nurse; serious mental illness
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This group will carry out the lifestyle intervention (Physical health promotion program) during 6 months.
  The group will attend a session per week.
  Interventions: Behavioral: Physical health promotion program
- Control group (No Intervention): usual care

INTERVENTIONS:
Behavioral: Physical health promotion program — The program has 24 sessions. Each session has two parts:
  * first part: half an hour of theoretical content, about the Metabolic syndrome, the effect of unhealthy lifestyle, toxic habits such as smoking or drinking alcohol, dietary habits or physical activity.
  * Second part: 1 hour of physical activity (walk)
  Arms: Experimental Group

SUMMARY:
The aim of this study is to evaluate the effectiveness of a lifestyle intervention, to reduce the risk of metabolic syndrome in patients with serious mental illness who receive treatment with antipsychotic medications.

The hypothesis of the study is that: the application of a physical health promotion program in people with serious mental illness, who receive treatment with antipsychotic medications, carried out by a mental health nurse, will decrease the presence of metabolic syndrome and contribute to improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of serious mental illness.
* Treatment with antipsychotics.
* Met at least 3 of the 5 criteria of metabolic syndrome According to the NCEP ATP III definition.

Exclusion Criteria:

* Medical contraindications to exercise
* Admitted to hospital.
* intellectual disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Decrease of at least 3 of the 5 criteria of metabolic syndrome | 6 months
  Fasting glucose ≥110 mg/dL (or receiving drug therapy for hyperglycemia) Blood pressure ≥130/85 mm Hg (or receiving drug therapy for hypertension) Triglycerides ≥150 mg/dL (or receiving drug therapy for hypertriglyceridemia) HDL-C <40 mg/dL in men or <50 mg/dL in women (or receiving drug therapy for reduced HDL-C) Waist circumference ≥102 cm in men or ≥88 cm in women

SECONDARY OUTCOMES:
Metabolic syndrome prevalence | 6 months
  expressed as a percentage
use of antipsychotic | 6 months
  Percentage of drugs prescribed by generic name
Toxic habits | 6 months
  Percentage of smokers percentage of people who drink alcohol percentage of people using drugs of abuse
Quality of life improvement | 6 months
  EuroQol- 5 Dimension (EQ-5D) includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).

CONTACTS AND LOCATIONS:
Locations (1):
- university hospital Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided